CLINICAL TRIAL: NCT02986321
Title: A 24-week, Multicenter, Randomized, Double-blind, Double-dummy, Placebo and Active Controlled, Parallel Group, Dose Ranging Study to Evaluate the Efficacy and Safety of 4 Doses of CHF6001 DPI in Patients With COPD on a Background Therapy
Brief Title: A 24-wk Dose Ranging Study to Evaluate the Efficacy and Safety of 4 Doses of a New PDE4 Inhibitor in Patients With COPD
Acronym: PIONEER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06001AA1-01; 2015-005548-32 (EudraCT Number)
Record Dates: First submitted 2016-11-24; First posted 2016-12-08 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: anti-inflammatory respiratory drug; PDE4 inhibitor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tanimilast; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CHF6001 DOSE1 (Experimental): DOSE1
  Interventions: Drug: CHF6001
- CHF6001 DOSE2 (Experimental): DOSE2
  Interventions: Drug: CHF6001
- CHF6001 DOSE3 (Experimental): DOSE3
  Interventions: Drug: CHF6001
- CHF6001 DOSE4 (Experimental): DOSE4
  Interventions: Drug: CHF6001
- Matched placebo (Placebo Comparator): placebo control
  Interventions: Drug: Placebo
- Budesonide (Active Comparator): Budesonide DPI 800µg
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: CHF6001 — Dose response: Test one of 4 different doses of CHF6001
  Other Names: Dose range finding
  Arms: CHF6001 DOSE1; CHF6001 DOSE2; CHF6001 DOSE3; CHF6001 DOSE4
Drug: Budesonide — active control
  Other Names: Active comparator
  Arms: Budesonide
Drug: Placebo — placebo control
  Arms: Matched placebo

SUMMARY:
The purpose of this study is to evaluate the dose-response relationship of different doses of CHF6001 and to identify the optimal dose (s) in terms of benefit/risk ratio for further development in the target patient population.

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blind, double-dummy, placebo and active controlled multinational, multicenter, dose ranging, 6-arm parallel-group study to identify the optimal dose of CHF6001, PDE4 inhibitor under development, with respect to lung functions and symptoms.

After a 2-wk run-in period under formoterol (Oxis Turbohaler®) and rescue salbutamol prn, patients will be randomized to one of the 6 treatment groups. After the randomization, patients will be assessed after 3, 6, 12, 18 and 24 weeks of treatment at clinic/hospital. A follow-up visit will be performed 12 days after the last visit.

During the study, patients will report daily symptoms with the EXACT-PRO/E-RS questionnaire, rescue/background medication use and compliance with the study medications. AEs, SAEs and COPD exacerbations will be monitored throughout the study. At randomization and subsequent visits, patients will undergo physical and vital signs examinations, spirometry measurement, 12-lead ECG. Symptoms and Health status will be assessed through validated questionnaires. Routine lab analysis and blood biomarkers will be done.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Non- childbearing potential or woman permanently sterilized or on one or more highly effective contraception
* Current/ex smokers (history > 10 pack years)
* Post bronchodilatator FEV1 >=30% and <=70% predicted normal value and FEV1/FVC ratio <0.7
* Documented history of at least 1 moderate or severe exacerbation in the 12 months prior to study entry
* Symptomatic patients (MMRC score ≥2 and a CAT score ≥10)
* Patients on daily maintenance therapy with an ICS/LABA .

Exclusion Criteria:

* Diagnosis of asthma or other respiratory disorders
* Maintenance bronchodilators therapy only (eg LABA alone)
* Maintenance triple therapy.
* Occurrence of a moderate or severe COPD exacerbation within 6 weeks prior to study entry or during the run-in period.
* Patients requiring long term oxygen therapy.
* Concomitant or recent pulmonary rehabilitation programme
* Known respiratory disorders other than COPD
* Lung cancer or a history of lung cancer, active or history of cancer with less than 5 years disease free survival time
* Hypersensitivity to β2-agonist, corticosteroids, PDE4 inhibitors or any of the excipients
* Depression, generalised anxiety disorder, suicidal ideation
* Any clinically significant cardiovascular disease (IM, CHF III/IV; AF not controlled by therapy, etc) within 1 year of study entry
* Any relevant clinically significant cardiovascular condition, clinically abnormal significant 12-lead ECG (QTcF>450 ms for male and >470 for female) or clinically significant laboratory abnormalities
* Serum potassium value ≤3.5 mEq/L or >5.5mEq/L and/or a fasting serum glucose value ≥140 mg/dL.
* History or symptoms of significant neurological disease
* Unstable concurrent disease: eg uncontrolled Thyroid disease or other endocrine diseases, gastrointestinal uncontrolled disease, uncontrolled immune diseases
* Renal impairment.
* Patients with abnormal alanine aminotransferase and/ or aspartate aminotransferase and/or bilirubin
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities and patients receiving treatment with any drug known to have a well defined potential for hepatotoxicity before Study entry
* Severely obese (BMI ≥35 kg/m2) or have experienced excessive weight loss recently
* History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening visit.
* Any recent participation to a clinical Study with other investigational drug

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in predose morning FEV1 at 12 weeks | week 12
  overall effect of CHF6001 on change from baseline in predose morning FEV1

SECONDARY OUTCOMES:
Change from baseline in predose morning FEV1 at other timepoints | weeks 3, 6, 18, 24
  Change from Baseline
Change from baseline in pre-dose morning IC | weeks 3, 6, 12, 18, 24
  Change from Baseline for other lung function parameters
Change from baseline in pre-dose morning FVC | weeks 3, 6, 12, 18, 24
  Change from Baseline for other lung function parameters
Change from baseline in TDI focal score | weeks 3, 6, 12, 18, 24
  Change of TDI score
Change from baseline in SGRQ score | weeks 3, 6, 12, 18, 24
  Change of SGRQ score
Change from baseline in E-RS score | weeks 3, 6, 12, 18, 24
  Change of E-RSI score
COPD exacerbation rate over 24 weeks of treatment | 24 weeks
  exacerbation rate
Time to first COPD exacerbation | 24 weeks
  Time to first COPD exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Principal Investigator — Medicines Evaluation Unit, Manchester, UK

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Govoni M, Bassi M, Santoro D, Donegan S, Singh D. Serum IL-8 as a Determinant of Response to Phosphodiesterase-4 Inhibition in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2023 Sep 1;208(5):559-569. doi: 10.1164/rccm.202301-0071OC. PMID 37192443
- [Derived] Singh D, Emirova A, Francisco C, Santoro D, Govoni M, Nandeuil MA. Efficacy and safety of CHF6001, a novel inhaled PDE4 inhibitor in COPD: the PIONEER study. Respir Res. 2020 Sep 22;21(1):246. doi: 10.1186/s12931-020-01512-y. PMID 32962709
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2015-005548-32